CLINICAL TRIAL: NCT03482180
Title: A Multi-Center, Randomized, Double-Blind, Parallel Phase III Study to Evaluate the Efficacy and Safety of KI1106 in Patients Whose TG Level is Not Adequately Controlled With Atorvastatin Calcium Monotherapy While LDL-C is Properly Controlled
Brief Title: Evaluate the Efficacy and Safety of KI1106 in Patients Whose TG Level is Not Adequately Controlled With Atorvastatin Calcium Monotherapy While LDL-C is Properly Controlled
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-OA-8301
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-03

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Group- KI1106 (Experimental): KI1106 tablet - daily administration
  Interventions: Drug: KI1106 4g, QD
- Control Group - Atorvastatin (Active Comparator): Atorvastatin Calcium 20mg - daily administration
  Interventions: Drug: Atorvastatin Calcium 20mg, QD

INTERVENTIONS:
Drug: KI1106 4g, QD — KI1106 4 Capsules
  Arms: Investigational Group- KI1106
Drug: Atorvastatin Calcium 20mg, QD — Atorvastatin Calcium 20mg
  Arms: Control Group - Atorvastatin

SUMMARY:
To examine variation rate of Non-HDL with KI1106 comparison Atorvastatin monotherapy.

DETAILED DESCRIPTION:
Randomly assigned to two groups (KI1106 or Atorvastatin monotherapy) after 4 weeks run-in period and prescribed KI1106 or Atorvastatin for 8 weeks.

ELIGIBILITY:
Inclusion criteria:

* Screening Visit

  * Age: 20-80
  * High risk for cardiovascular disease according to NCEP APT III
  * TG≥300mg/dL and 160mg/dL>LDL-C≥100mg/dL for subjects who were not taking statins for 4 weeks
  * 500mg/dL>TG≥200mg/dL and LDL-C<110mg/dL for subjects who were taking statins for 4 weeks
* Baseline Visit

  * 500mg/dL>TG≥200mg/dL
  * LDL-C<110mg/dL
  * Reduction of LDL-C comparing screening visit

Exclusion criteria:

* The patient has histories of acute artery disease within 3 months
* The patient has histories of operation revasculariation or aneurysm within 6 months
* The patient has histories of unexplained myalgia or diagnosed myalgia or rhabdomyolysis
* The patient has histories of effect able disease to the procedure and clinical trial result

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Variation rate of Non HDL-C | 8 weeks

SECONDARY OUTCOMES:
Variation rate of TG | 4 weeks, 8 weeks
Variation rate of Non HDL-C | 4 weeks
Variation rate of TC | 4 weeks, 8 weeks
Variation rate of LDL-C | 4 weeks, 8 weeks
Variation rate of VLDL-C | 4 weeks, 8 weeks
Variation rate of Apo A-I | 4 weeks, 8 weeks
Variation rate of Apo B | 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: kyungshun Shin, Dr, Study Director — manager

IPD SHARING:
Plan to Share IPD: No